CLINICAL TRIAL: NCT06098274
Title: The Effect of Transtheoretic Model and Motivational Interview Based Intervention Program on Smartphone Addiction and Sleep Quality Levels in Nursing Students
Brief Title: Motivational Interview Based Intervention Program on Smartphone Addiction and Sleep Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mustafa Yumusak (Other)
Collaborators: Cumhuriyet University (Other)
Responsible Party: Sponsor-Investigator, Mustafa Yumusak, Research assistant, Aksaray University
Organization: Aksaray University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AksarayUniversity
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Smartphone Addiction; Students, Nursing
Keywords: smartphone addiction; sleep quality; motivational interview; transtheoretical model; nursing student
MeSH Terms: conditions — Internet Addiction Disorder; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The method of this research; It is a quasi-experimental study with pre-test and post-test, with intervention and control groups randomly selected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing group based on transtheoretical model (Experimental): Smartphone addiction scale will be applied to nursing department students. Those who score 31 or more on the scale for men and 33 or more for women will be considered at risk and will be invited to the study. Those who meet the participation criteria and volunteer to participate will be included in the study. Participants will be homogeneously and randomly distributed into intervention and control groups.
  Interventions: Behavioral: Motivational interviewing program based on transtheoretical model
- Group without transtheoretical model-based motivational interviewing (Control group) (No Intervention): No intervention will be made to the intervention group. After evaluating the final data, if the motivational interview and training program is found to be effective, a motivational interview and training program will also be carried out to the control group participants.

INTERVENTIONS:
Behavioral: Motivational interviewing program based on transtheoretical model — It will be determined at which stage of change of the transtheoretic model the participants in the intervention group are. A varying number of motivational interviews will be held depending on the stage of change and a maximum of 6 motivational interviews. Those in the preparatory phase will be trained on smartphone addiction. Following completion of the motivational interviewing and training content, the study scales will be re-administered and the effectiveness of the motivational interviewing and training content will be evaluated by comparison with the baseline data.
  Arms: Motivational interviewing group based on transtheoretical model

SUMMARY:
Smartphones are the technological devices of our age that are constantly evolving and whose use is becoming more widespread day by day. Smartphones, which are preferred by almost everyone for reasons such as being easily portable, providing quick access to transactions, providing ease of use and sometimes as a status indicator, can pose a risk of addiction when used uncontrolled. Since young people are more intertwined with technology and use smartphones more, they are at greater risk of addiction and the problems that addiction can cause. Poor sleep quality is an important problem that can occur with smartphone addiction and negatively affects both daily life and the health of the individual. Smartphone addiction and the problems it causes are an important public health problem that threatens the whole society, especially young people. In solving this problem, it is among the duties of nurses to teach individuals healthy lifestyle behaviors instead of problematic behaviors. A road map is needed to facilitate the behavior change process. Transtheoretical Model (TTM) is widely used today to improve the behavior change process in the individual and to achieve the most effective health behavior change. TTM, which targets interventions appropriate to the individual's stage of change, is used as a guide that facilitates behavioral change. TTM is a model that contributes to change, accelerates it, and supports individuals considering change. In addition to TTM, another method that is more frequently used and contributes to change, especially in addicted individuals, is the "motivational interviewing" method. Motivational interviewing is very effective in gaining positive health behaviors and changing negative health behaviors and aims to reveal the individual's internal motivation. It is thought that the university years, which are an important period in terms of developing and maintaining health-protective and preventive behaviors, will both increase students' health responsibility and protect them from health-threatening behaviors with the healthy lifestyle behaviors acquired during this period. In line with all this information, this study was planned to determine the effect of the Transtheoretical model and motivational interview-based online intervention program on smartphone addiction and sleep quality levels in nursing students who are in the smartphone addiction risk group.

DETAILED DESCRIPTION:
Smartphones are the technological devices of our age that are constantly developing and their use is becoming more widespread every day. Nowadays, many transactions from shopping to banking activities, playing mobile games and taking photos can be done easily with smart phones. Smart phones, which make positive contributions to daily life, attract great attention by individuals of all age groups, especially young people. According to Newzoo's report, the number of smartphone users, which was 3.5 billion in 2020, is expected to reach 4.1 billion in 2023. Smartphones, which are preferred by almost everyone for reasons such as being easily portable, providing fast access in transactions, ease of use and sometimes a status indicator, can pose a risk for addiction when used uncontrolled. Smartphone addiction, although not yet clearly defined; It can manifest itself with symptoms such as constantly checking the phone, feeling restless when staying away, withdrawing, mood changes, not being able to control the duration of use, disruption in daily life due to problematic use, constant desire to use and pleasure from use. According to the behavioral approach, if a person takes pleasure from a behavior or avoids negative emotions with this behavior, this situation turns into a habit in the individual. Uncontrollable and frequently repetitive habits carry a risk for addiction. Smartphone addiction, in addition to being a behavioral disorder, can cause many physical, social and psychological problems. Problematic use of the smartphone; decrease in sleep duration and quality, height, wrist, thumb and shoulder pain , dry eye syndrome, and eye fatigue, decreased physical activity, as well as depression, social phobia, loneliness, and decreased academic performance can bring along many psychological and social problems. It can be said that poor sleep quality is one of the primary problems that may occur in the problematic use of the smartphone, and it negatively affects both daily life and the health of the individual. Especially at night and in the pre-sleep period, the use of smartphones adversely affects sleep quality as it causes arousal due to the blue light it emits, shortens the sleep duration and disrupts the circadian rhythm. A study stated that exposure to blue light 1 hour before sleep reduces the duration of deep sleep and causes sleep quality to deteriorate. Another study stated that leaving smartphones out of the bedroom improved sleep quality. It is stated that poor sleep quality negatively affects the individual physically and psychologically, causes performance losses and increases the risk of accidents. In studies conducted with students, it was stated that poor sleep quality negatively affects academic performance, while good sleep quality increases academic performance. A study conducted with adolescents stated that poor sleep quality was associated with low self-esteem and increased levels of anxiety and depression. Nurses, who serve almost all of the society, have an important role in defining risky health behaviors and planning and implementing appropriate interventions for behavior change. For this reason, nurses need to make an effort to find the most appropriate behavior change approaches for the individual. Today, the Transtheoretic Model (TTM) is widely used to improve the behavior change process in the individual and to achieve the most effective health behavior change. TTM, which aims at the initiative suitable for the change phase of the individual, is used as a guide that facilitates behavior change. TTM is a cognitive-behavioral model that accepts that any behavioral change in an individual does not happen all at once, but that behavior change includes different stages and processes. The model, which was first used in smoking cessation programs, was later used in many areas such as exercise, sun protection, reducing the amount of excess fat in the diet, weight control, condom use, supporting mammography screening, widespread drug use, coping with stress and quitting substance abuse. Traditional behavior change models have an understanding that does not take into account the change stage of the individual or accepts that all individuals have the same level of readiness for behavior change. it is stated that the initiatives applied without considering the individual's readiness level for behavior change develop resistance to behavior change. In TTM, behavior change; It is defined as a gradual, continuous and dynamic structure. Change in traditional behaviorist approaches; In this model, change focuses on helping individuals willingly make behavioral change and understanding the change process. In other words, it does not classify individuals only according to whether they can perform a certain behavior, but also according to the stages passed in the behavior change process. While TTM creates a roadmap in change, there are also approaches that contribute to and accelerate this change and support the individual who thinks about change. One of these approaches, which is used more frequently in addicted individuals, is the "motivational interview" method. Motivational interviewing is very effective in gaining positive health behaviors and changing negative health behaviors and can be an effective communication technique for nurses in providing behavior change. Motivational interviewing as defined by Miller; "It is a client-centered interview form in which suggestions are made to provide behavior change by helping individuals discover and solve their problems". In motivational interviewing, the expert is the consultant, but the consultant does not assume the role of the knower, is not ready before the client, does not impose his own thoughts, wherever the client is, the consultant is directed there. Solving problems in motivational interviewing is the client's job, not the counselor's. Direct persuasion, aggressive confrontation and discussion are the conceptual opposites of motivational interviewing. Motivational interviewing is accompaniment and non-judgmental acceptance. In the interview, the energy of the client should be used and his desire for change should be revealed. motivational interview; It is a partnership-friendship relationship rather than an expert-recipient role. The counselor should respect the client's autonomy, freedom to make choices and bear the consequences. Nurses, who have very important roles and duties in the provision of health services to the society, undertake important duties not only at the point of care for the sick individual, but also in the fight against situations that threaten public health. In particular, public health nurses interact not only with patients but also with the entire society they serve, as they work in primary health care institutions. Smartphone addiction and the problems it causes are an important public health problem that threatens the whole society and especially young individuals. In the solution of this problem, it is also among the duties of the public health nurse to provide the individual with healthy lifestyle behaviors instead of problematic behavior. As in all risky behaviors that threaten public health, the public health nurse provides consultancy services to the society as a requirement of education and consultancy in smart phone addiction and informs the society about the problems that may arise with the trainings it will organize. Based on this information, the reason for the selection of nursing students in the research universe; To raise awareness among students and contribute to public health, since nursing students are candidates to provide health services to the society, they are role models for the society with their healthy lifestyle behaviors, they interact with individuals from all parts of the society in business life, and there are institutions that provide service on addiction among their work areas. decided with consideration. Another important factor in the selection of the research population is that, considering smartphone addiction, especially young individuals are more at risk for addiction and the problems that may arise from addiction, as they are more intertwined with technology and use smartphones more. According to the data of the Turkish Statistical Institute (TUIK) for 2021, it is stated that the rate of smartphone usage is higher for people with a university level education. In studies conducted in our country and abroad, approximately 50% of university students expressed themselves as smartphone addicts. Considering that being away from family and being more active in social life increases the need for communication among university students, it can be said that they are at higher risk for smartphone addiction when it is considered that they are not under family supervision since most of them reside in dormitories or student houses. In studies evaluating the smart phone usage habits of university students; It has been concluded that they use it for 6 hours or more, the purpose of their use is communication and access to social media, they use it more intensively in the evening and late at night, and they always keep it with them in the pre-sleep period. In studies examining the results of smartphone addiction in university students, results such as decrease in sleep quality, decrease in academic performance, depression, anxiety, muscle and joint pain were reached. It is thought that the university years, which are an important period for the development and maintenance of health protective and preventive behaviors, will both increase the health responsibility of the students and protect them from health-threatening behaviors with the healthy lifestyle behaviors to be gained in this period. It is seen that studies on smartphone addiction are generally descriptive studies aimed at determining the situation. Almost all of the intervention studies that could be reached were carried out in Far East countries and different intervention methods were used. In intervention studies aimed at preventing smartphone addiction; motivational interviewing, cognitive behavioral therapy, laughter therapy, sand play therapy, literacy therapy, peer relations development program, music therapy , mind-bending meditation program, mind-body exercise, journaling, and art therapy have been reached. In line with all this information, our study was planned to determine the effect of TTM and motivational interview-based online intervention program on smartphone addiction and sleep quality levels in nursing students who are in the risk group for smartphone addiction.

ELIGIBILITY:
Inclusion Criteria:

* Aksaray University Faculty of Health Sciences, Nursing Department 1st, 2nd, 3rd and 4th year students
* Those who have been using smartphones for at least 1 year
* Those who score above the cut-off score on the Smartphone Addiction Scale-Short Form (31 for men, 33 for women)
* Those who do not have internet access problems
* Those who volunteer to participate in the study and have no problems communicating

Exclusion Criteria:

* Having a chronic disease, diagnosed psychiatric health problem or sleep problem
* The individual does not want to continue working or does not attend a maximum of 2 motivational interview sessions.
* Having to take a break from education or terminate university education

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | 1. week
  The form, which was created to determine students' socio-demographic characteristics and smartphone usage habits, was prepared by the researcher in line with the literature review on the subject. The form consists of a total of 18 questions; There are 8 questions about the socio-demographic characteristics of the students, 8 questions evaluating smartphone usage characteristics, and 2 questions evaluating the individual's smartphone addiction and sleep quality by self-report.
Smartphone Addiction Scale Short Form (SAS-SF) | 1. week
  The scale is a 6-point Likert type and consists of 10 items. The lowest score from the scale can be 10 and the highest score can be 60. Increasing the total score from the scale indicates that the risk for smartphone addiction increases. The cut-off score of the scale in the Korean sample was determined as 31 for men and 33 for women.
Pittsburgh Sleep Quality Index (PSQI) | 1. week
  Pittsburgh Sleep Quality Index consists of 18 questions in which the individual evaluates himself. The scale consists of 7 components in total. These; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime sleep dysfunction. Each component is evaluated separately on a scale of 0-3 points. The total score that can be obtained from the Pittsburgh Sleep Quality Index varies between 0-21. A total score of 5 or less on the scale is interpreted as "good" sleep quality, and a score above 5 is interpreted as "bad" sleep quality.
Classification of Stages of Change Scale | 1. week
  The Stages of Change Classification Scale indicates the stages of change that individuals go through when they try to change their problematic behavior alone or with support. The stages of change that the individual goes through were developed based on the Transtheoretic Model. The scale guides the practices necessary for the individual to move on to the next stage of change. There is no scoring on the scale, and participants are divided into stages based on their answers to the questions.
  1. Not Considering Change Stage: It is the stage where behavior change is not considered.
  2. Consideration Stage: This is the stage where behavior change is considered within the next six months.
  3. Preparation Phase: This is the phase where behavioral change is considered within the next month.
  4. Action Phase: This is the phase where behavioral change begins to be implemented.
  5. Maintenance Phase: This is the phase that covers six months and indefinite period following the behavioral change.

SECONDARY OUTCOMES:
Smartphone Addiction Scale Short Form (SAS-SF) | 16. week
  The scale is a 6-point Likert type and consists of 10 items. The lowest score from the scale can be 10 and the highest score can be 60. Increasing the total score from the scale indicates that the risk for smartphone addiction increases. The cut-off score of the scale in the Korean sample was determined as 31 for men and 33 for women.
Pittsburgh Sleep Quality Index (PSQI) | 16. week
  Pittsburgh Sleep Quality Index consists of 18 questions in which the individual evaluates himself. The scale consists of 7 components in total. These; subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime sleep dysfunction. Each component is evaluated separately on a scale of 0-3 points. The total score that can be obtained from the Pittsburgh Sleep Quality Index varies between 0-21. A total score of 5 or less on the scale is interpreted as "good" sleep quality, and a score above 5 is interpreted as "bad" sleep quality.
Classification of Stages of Change Scale | 16. week
  The Stages of Change Classification Scale indicates the stages of change that individuals go through when they try to change their problematic behavior alone or with support. The stages of change that the individual goes through were developed based on the Transtheoretic Model. The scale guides the practices necessary for the individual to move on to the next stage of change. There is no scoring on the scale, and participants are divided into stages based on their answers to the questions.
  1. Not Considering Change Stage: It is the stage where behavior change is not considered.
  2. Consideration Stage: This is the stage where behavior change is considered within the next six months.
  3. Preparation Phase: This is the phase where behavioral change is considered within the next month.
  4. Action Phase: This is the phase where behavioral change begins to be implemented.
  5. Maintenance Phase: This is the phase that covers six months and indefinite period following the behavioral change.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Yumuşak, Principal Investigator — Aksaray University; Semra Kocataş, Study Director — Cumhuriyet University
Locations (2):
- Turkey (Türkiye) (2):
  - Aksaray University, Aksaray
  - Sivas Cumhuriyet University, Sivas

IPD SHARING:
Plan to Share IPD: Yes
Sociodemographic data of participants, Smartphone Addiction Scale Short Form results, Pittsburgh Sleep Quality Index results, Classification of Stages of Change Scale results
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: The Council of Higher Education will be shared from the thesis center.
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/

REFERENCES:
- [Background] Newzoo Global Mobile Market Report 2020, Free Version. Available online: https://newzoo.com/insights/trend-reports/newzoo-global-mobile-market-report-2020-free-version/ (Date of access: 19.10.2023).
- [Background] Li L, Lin TTC. Over-connected? A qualitative exploration of smartphone addiction among working adults in China. BMC Psychiatry. 2019 Jun 18;19(1):186. doi: 10.1186/s12888-019-2170-z. PMID 31215473
- [Background] Mohamed SM, Mostafa MH. Impact of smartphone addiction on depression and self-esteem among nursing students. Nurs Open. 2020 May 19;7(5):1346-1353. doi: 10.1002/nop2.506. eCollection 2020 Sep. PMID 32802355
- [Background] Oulasvirta, A., Rattenbury, T., Ma, L., & Raita, E. (2012). Habits make smartphone use more pervasive. Personal and Ubiquitous Computing, 16(1), 105-114.
- [Background] Grant JE, Potenza MN, Weinstein A, Gorelick DA. Introduction to behavioral addictions. Am J Drug Alcohol Abuse. 2010 Sep;36(5):233-41. doi: 10.3109/00952990.2010.491884. PMID 20560821
- [Background] Randler C, Wolfgang L, Matt K, Demirhan E, Horzum MB, Besoluk S. Smartphone addiction proneness in relation to sleep and morningness-eveningness in German adolescents. J Behav Addict. 2016 Sep;5(3):465-73. doi: 10.1556/2006.5.2016.056. Epub 2016 Aug 8. PMID 27499228
- [Background] Amez S, Vujic S, Soffers P, Baert S. Yawning while scrolling? Examining gender differences in the association between smartphone use and sleep quality. J Sleep Res. 2020 Dec;29(6):e12971. doi: 10.1111/jsr.12971. Epub 2020 Jan 9. PMID 31919946
- [Background] AlAbdulwahab SS, Kachanathu SJ, AlMotairi MS. Smartphone use addiction can cause neck disability. Musculoskeletal Care. 2017 Mar;15(1):10-12. doi: 10.1002/msc.1170. Epub 2017 Jan 19. No abstract available. PMID 28105706
- [Background] Choi, Y. S. (2018). A study on the smartphone addiction and physical pain in the university students. Biomed Res, 29, 3162-8.
- [Background] Baabdullah A, Bokhary D, Kabli Y, Saggaf O, Daiwali M, Hamdi A. The association between smartphone addiction and thumb/wrist pain: A cross-sectional study. Medicine (Baltimore). 2020 Mar;99(10):e19124. doi: 10.1097/MD.0000000000019124. PMID 32150053
- [Background] Xie Y, Szeto GP, Dai J, Madeleine P. A comparison of muscle activity in using touchscreen smartphone among young people with and without chronic neck-shoulder pain. Ergonomics. 2016;59(1):61-72. doi: 10.1080/00140139.2015.1056237. Epub 2015 Jul 28. PMID 26218600
- [Background] Paek, K. S. (2017). A convergence study the association between addictive smart phone use, dry eye syndrome, upper extremity pain and depression among college students. Journal of the Korea Convergence Society, 8(1), 61-69.
- [Background] Golebiowski B, Long J, Harrison K, Lee A, Chidi-Egboka N, Asper L. Smartphone Use and Effects on Tear Film, Blinking and Binocular Vision. Curr Eye Res. 2020 Apr;45(4):428-434. doi: 10.1080/02713683.2019.1663542. Epub 2019 Oct 7. PMID 31573824
- [Background] Haripriya, S., Samuel, S. E., & Megha, M. (2019). Correlation between Smartphone Addiction, Sleep Quality and Physical Activity among Young Adults. Journal of Clinical & Diagnostic Research, 13(10).
- [Background] Alhassan AA, Alqadhib EM, Taha NW, Alahmari RA, Salam M, Almutairi AF. The relationship between addiction to smartphone usage and depression among adults: a cross sectional study. BMC Psychiatry. 2018 May 25;18(1):148. doi: 10.1186/s12888-018-1745-4. PMID 29801442
- [Background] Hawi, N. S., & Samaha, M. (2017). Relationships among smartphone addiction, anxiety, and family relations. Behaviour & Information Technology, 36(10), 1046-1052.
- [Background] Enez Darcin, A., Kose, S., Noyan, C. O., Nurmedov, S., Yılmaz, O., & Dilbaz, N. (2016). Smartphone addiction and its relationship with social anxiety and loneliness. Behaviour & Information Technology, 35(7), 520-525.
- [Background] Baert, S., Vujić, S., Amez, S., Claeskens, M., Daman, T., Maeckelberghe, A., Omey, E., and De Marez, L. (2020) Smartphone Use and Academic Performance: Correlation or Causal Relationship?. Kyklos, 73: 22- 46. https://doi.org/10.1111/kykl.12214
- [Background] Jniene A, Errguig L, El Hangouche AJ, Rkain H, Aboudrar S, El Ftouh M, Dakka T. Perception of Sleep Disturbances due to Bedtime Use of Blue Light-Emitting Devices and Its Impact on Habits and Sleep Quality among Young Medical Students. Biomed Res Int. 2019 Dec 24;2019:7012350. doi: 10.1155/2019/7012350. eCollection 2019. PMID 31950050
- [Background] Ishizawa M, Uchiumi T, Takahata M, Yamaki M, Sato T. Effects of pre-bedtime blue-light exposure on ratio of deep sleep in healthy young men. Sleep Med. 2021 Aug;84:303-307. doi: 10.1016/j.sleep.2021.05.046. Epub 2021 Jun 8. PMID 34217920
- [Background] Hughes, N., & Burke, J. (2018). Sleeping with the frenemy: How restricting 'bedroom use'of smartphones impacts happiness and wellbeing. Computers in Human Behavior, 85, 236-244.
- [Background] Watson NF, Badr MS, Belenky G, Bliwise DL, Buxton OM, Buysse D, Dinges DF, Gangwisch J, Grandner MA, Kushida C, Malhotra RK, Martin JL, Patel SR, Quan SF, Tasali E. Recommended Amount of Sleep for a Healthy Adult: A Joint Consensus Statement of the American Academy of Sleep Medicine and Sleep Research Society. Sleep. 2015 Jun 1;38(6):843-4. doi: 10.5665/sleep.4716. PMID 26039963
- [Background] El Hangouche AJ, Jniene A, Aboudrar S, Errguig L, Rkain H, Cherti M, Dakka T. Relationship between poor quality sleep, excessive daytime sleepiness and low academic performance in medical students. Adv Med Educ Pract. 2018 Sep 7;9:631-638. doi: 10.2147/AMEP.S162350. eCollection 2018. PMID 30233270
- [Background] Adelantado-Renau M, Diez-Fernandez A, Beltran-Valls MR, Soriano-Maldonado A, Moliner-Urdiales D. The effect of sleep quality on academic performance is mediated by Internet use time: DADOS study. J Pediatr (Rio J). 2019 Jul-Aug;95(4):410-418. doi: 10.1016/j.jped.2018.03.006. Epub 2018 May 19. PMID 29787701
- [Background] Woods HC, Scott H. #Sleepyteens: Social media use in adolescence is associated with poor sleep quality, anxiety, depression and low self-esteem. J Adolesc. 2016 Aug;51:41-9. doi: 10.1016/j.adolescence.2016.05.008. Epub 2016 Jun 10. PMID 27294324
- [Background] Erol, S., & Erdoğan, S. (2007). Sağlık davranışlarını geliştirmek ve değiştirmek için transteoratik modelin kullanılması. Atatürk Üniversitesi Hemşirelik Yüksekokulu Dergisi, 10(2), 86-94.
- [Background] Taş, F., Seviğ, E. Ü., Güngörmüş, Z. (2016). Sigara bağımlılığında davranış değişimi için transteoretik model ile motivasyonel görüşme tekniğinin kullanılması. Psikiyatride Güncel Yaklaşımlar, 8(4), 380-392.
- [Background] Güngörmüş Z (2010) Lise öğrencilerinde sigara içme davranışının Transteoretik model çerçevesinde değerlendirilmesi. Sürekli Tıp Eğitimi Dergisi, 19:12-18.
- [Background] Sertel HÖ, Yücel B, Deveci E. ergenlik döneminde obezite; bilişsel davranışçı kuramlar ve motivasyon kuramları açısından karşılaştırmalı bir inceleme, Türkiye Klinikleri J Psychol-Special Topics, 2016;1(2):50-58.
- [Background] Walters JA, Courtney-Pratt H, Cameron-Tucker H, Nelson M, Robinson A, Scott J, Turner P, Walters EH, Wood-Baker R. Engaging general practice nurses in chronic disease self-management support in Australia: insights from a controlled trial in chronic obstructive pulmonary disease. Aust J Prim Health. 2012;18(1):74-9. doi: 10.1071/PY10072. PMID 22394666
- [Background] Rollnick S, Miller WR. What is motivational in-terviewing? Behav Cognit Psychother 1995; 23(4):325- 34.
- [Background] Ögel K. Motivasyonel görüşme tekniği. Türkiye Klinikleri Psychiatry-Special Topics 2009; 2(2):41- 4.
- [Background] Augner C, Hacker GW. Associations between problematic mobile phone use and psychological parameters in young adults. Int J Public Health. 2012 Apr;57(2):437-41. doi: 10.1007/s00038-011-0234-z. Epub 2011 Feb 3. PMID 21290162
- [Background] Cocoradă, E., Maican, C. I., Cazan, A. M., & Maican, M. A. (2018). Assessing the smartphone addiction risk and its associations with personality traits among adolescents. Children and Youth Services Review, 93, 345-354.
- [Background] TÜİK (2021), Hanelerde Bilişim Teknolojileri Kullanım Araştırması, https://data.tuik.gov.tr/Bulten/Index?p=Hanehalki-Bilisim-Teknolojileri-(BT)-Kullanim-Arastirmasi-2021-37437 , (Date of access; 18.10.2023).
- [Background] Aljomaa, S. S., Qudah, M. F. A., Albursan, I. S., Bakhiet, S. F., & Abduljabbar, A. S. (2016). Smartphone addiction among university students in the light of some variables. Computers in Human Behavior, 61, 155-164.
- [Background] Ghosh T, Sarkar D, Sarkar K, Dalai CK, Ghosal A. A study on smartphone addiction and its effects on sleep quality among nursing students in a municipality town of West Bengal. J Family Med Prim Care. 2021 Jan;10(1):378-386. doi: 10.4103/jfmpc.jfmpc_1657_20. Epub 2021 Jan 30. PMID 34017757
- [Background] Wang PY, Chen KL, Yang SY, Lin PH. Relationship of sleep quality, smartphone dependence, and health-related behaviors in female junior college students. PLoS One. 2019 Apr 3;14(4):e0214769. doi: 10.1371/journal.pone.0214769. eCollection 2019. PMID 30943270
- [Background] Yumuşak M., (2019). Üniversite öğrencilerinde akıllı telefon bağımlılığı, uyku kalitesi ve yaşam doyumu düzeyleri, Yükseklisans Tezi, Erciyes Üniversitesi Sağlık Bilimleri Enstitüsü, Kayseri, 33-34.
- [Background] Setiawan, A., Sugiharto, D. Y. P., & Purwanto, E. (2021). Efektivitas Konseling Motivational Interviewing (MI) dalam Mereduksi Adiksi Smartphone Siswa. In Prosiding Seminar Nasional Bimbingan dan Konseling Universitas Ahmad Dahlan (Vol. 1).
- [Background] Khalily MT, Bhatti MM, Ahmad I, Saleem T, Hallahan B, Ali SA, Khan AA, Hussain B. Indigenously adapted cognitive-behavioral therapy for excessive smartphone use (IACBT-ESU): A randomized controlled trial. Psychol Addict Behav. 2021 Feb;35(1):93-101. doi: 10.1037/adb0000677. Epub 2020 Jul 23. PMID 32700919
- [Background] Lu, C., Zou, L., Becker, B., Griffiths, M. D., Yu, Q., Chen, S. T., ... & Zhang, Y. (2020). Comparative effectiveness of mind-body exercise versus cognitive behavioral therapy for college students with problematic smartphone use: a randomized controlled trial. International Journal of Mental Health Promotion, 22(4), 271-282.
- [Background] Shin, J. H., & Jang, M. (2016). Effect of group sandplay therapy to be addicted youth's addiction levels and anxiety. Journal of Symbols & Sandplay Therapy, 7(1), 39-55.
- [Background] Baek, H. G., & Ha, T. H. (2018). A Study on the Effects of Literacy Therapy Program for the Prevention of Adolescents' Smartphone Addiction. Journal of Digital Contents Society, 19(2), 269-276.
- [Background] Bong SH, Won GH, Choi TY. Effects of Cognitive-Behavioral Therapy Based Music Therapy in Korean Adolescents with Smartphone and Internet Addiction. Psychiatry Investig. 2021 Feb;18(2):110-117. doi: 10.30773/pi.2020.0155. Epub 2021 Feb 2. PMID 33517616
- [Background] Jo J, Bang KS. The effect of peer relationship enhancement programs on the prevention of smartphone addiction among late school-age children in South Korea. J Pediatr Nurs. 2022 Mar-Apr;63:e127-e135. doi: 10.1016/j.pedn.2021.09.025. Epub 2021 Oct 5. PMID 34625302
- [Background] Yoo, Y. G., Lee, M. J., Yu, B., & Yun, M. R. (2019). The effect of Mind Subtraction Meditation on smartphone addiction in school children. Glob. J. Health Sci, 11, 16-28.
- [Background] Lee H, Seo MJ, Choi TY. The Effect of Home-based Daily Journal Writing in Korean Adolescents with Smartphone Addiction. J Korean Med Sci. 2016 May;31(5):764-9. doi: 10.3346/jkms.2016.31.5.764. Epub 2016 Mar 23. PMID 27134499
- [Background] Jang, H. J., Kim, J. W., & Choi, T. Y. (2017). The effect of group therapy using art program on Internet/Smartphone addictive behaviors of adolescents: a pilot study. J Korean Soc Biol Ther Psychiatry, 23, 171-180.
- [Background] Bae, S. Y., & Won, H. R. (2019). The effect of attachment-focused group art therapy on early youth attachment behavior and smartphone overdependence. Korean J. Arts Ther, 26, 559-584.
- [Background] Choi, W., Park, J., Jung, H., Yim, J., Lee, S., Han, S., Park, S., Jeong, H. (2016). The effects of laughter therapy interventions for smartphone addicts. International Journal of Bio-Science and Bio-Technology, 8(4), 189-198.
- [Background] Choi EH, Chun MY, Lee I, Yoo YG, Kim MJ. The Effect of Mind Subtraction Meditation Intervention on Smartphone Addiction and the Psychological Wellbeing among Adolescents. Int J Environ Res Public Health. 2020 May 7;17(9):3263. doi: 10.3390/ijerph17093263. PMID 32392863